CLINICAL TRIAL: NCT05785000
Title: Rehabilitation of Adult Patients With Post Concussion Syndrome
Brief Title: Rehabilitation in Post Concussion Syndrome
Acronym: REPCon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University College Copenhagen (Other)
Responsible Party: Principal Investigator, Henrik Bo Wiberg Larsson, Consultant, professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Repcon123
Record Dates: First submitted 2023-03-06; First posted 2023-03-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-04

CONDITIONS: Post-Concussion Syndrome
Keywords: Mild traumatic brain injury; Brain function; Magnetic Resonance Imaging; Buffalo Concussion Bike Test; Patient perception; 360-degree evaluation
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion

STUDY DESIGN:
Intervention Model Description: Patients are recruited through our professional networks, via clinics, hospital emergency departments, general practitioners, physiotherapeutic clinics, flyers at educational institutions and patient associations. Inclusion age is 18-70 years, both genders. PCS symptoms of at least 4 weeks persistence after initial trauma and patients must be able to document the traumatic brain event from either emergency room or other medical doctor. Exclusion criteria: other diseases interfering with presentation of PCS symptoms.
  Up to fifty healthy controls are included only in the MRI part. Healthy controls are recruited by advertising in public media. This part of the project is also constituted as a separate case control study comparing PCS patients and healthy controls
  Seventy patients with PCS are randomized to either intervention as an add on to usual care or to control. Randomization is performed as a block-randomization with permuted block of size 2-6 generated via computer.
Who Masked: Outcomes Assessor
Masking Description: The assessors of outcomes at the end of the project are different to the assessors of clinical test at entry to the project
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobe graded physical exercise intervention and usual care (Experimental): Physical exercise program. The experimental programme is an add-on to usual care and consists of an aerobe graded exercise program performed twice a week for 12 weeks. Usual care includes all public treatments that each patient is assigned to at entry to REPCon. The provision of officially available treatments follow the Danish Health Care Act.
  Interventions: Other: Physical exercise programme as an add-on
- Usual care (Placebo Comparator): No physical exercise program in a patient control group with PCS. This group continues with usual care, but all clinical test, interviews and MRI protocol are the same.
  Interventions: Other: Control patients receiving usual care

INTERVENTIONS:
Other: Physical exercise programme as an add-on — Consists of an individually tailored bike exercise program guided by symptoms, pulse rate and patient specific judgement of exertion monitored also by BORG RPE and VAS and progressively increasing time and level of resistance below symptom provocation
  Arms: Aerobe graded physical exercise intervention and usual care
Other: Control patients receiving usual care — No exercise intervention
  Arms: Usual care

SUMMARY:
This project evaluates and quantifies the effects of an individually tailored exercise program applied to patients with long-lasting symptoms after concussion, minor traumatic brain injury, so-called Post-Concussion Syndrome (PCS). The project investigates the phenomenon Post Concussion Syndrome in four dimensions with a focus on both patient perspectives of PCS, an interventional physical program, a neurobiological basis for PCS through Magnetic Resonance Imaging (MRI) and finally through a 360-degree evaluation of the entire project involving patients and scientists in a reflective process.

DETAILED DESCRIPTION:
The project has four parts

Aims and hypotheses:

1. The aim is to describe and nuance the subjective patient perceived aspects of living with PCS including the individual experiences of symptom provocation or relieve after the initial trauma. Part one is concept developing and involves qualitative in-depth interviews of patient experiences of obstacles for living a normal life with special emphasis of intolerance to activity and exercise.
2. The aim is to assess the effects of adding a 12 week individually tailored pulse-controlled aerobe exercise program to usual care. The hypothesis is that it is possible to increase the physical capacity measured by the number of minutes of pulse-training without symptom provocation. By increasing the number of minutes the threshold value of symptom provocation will be moved upwards for a training group (TG) of patients compared to a control group (CG) who carry on in their usual activities and treatments here defined as usual care.
3. The aim is to measure quantitative components of the neurobiological aspects of PCS by magnetic resonance imaging (MRI). The hypothesis is that patients with PCS have more leakiness of the blood-brain barrier (BBB) compared to healthy controls. In addition, PCS patients have disturbance of brain metabolism, abnormal microstructural tissue organization and abnormal brain activity. Furthermore, that intervention will normalize these MRI metrics in a training group (TG) compared to a control group (CG).
4. The aim is to obtain qualitative components of having patients and scientists evaluating the project. The evaluation will comprise participants involved, i.e. both patients in the 2 arms and researchers and the goal of this 360-degree evaluation is to describe perceived experiences of strength, weakness, possibility and threat (SWOT) of the intervention and ultimately prevent development of PSC after a minor traumatic brain injury.

Methods - the four parts:

1. Qualitative interviews of PCS participants focusing on individual perception of own situation, detailed symptom description, hindrance of living a normal life.
2. All PSC patients continue daily living and own developed coping strategies. The intervention is an add-on. We use Short Message Service (SMS) tracking every week obtaining details of wellbeing related to living with concussion. The intervention consists of bi-weekly one hour exercise guided by physiotherapist for 12 weeks. Clinical status is performed four times- before and after 12 weeks and with two interim assessments. We use the validated Buffalo Concussion Bike Test (BCBT ). Blood pressure, pulse rate, pulse oxymetri and exercise level are registered and we use Visual Analog Scale (VAS) and BORG Ratings of Perceived Exertion (BORG RPE) scales. In addition we use the Rivermead Post Concussion Questionnaire (RPCQ ).
3. Blood brain barrier (BBB) permeability is measured by Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE-MRI) using a conventional MRI contrast agent. Both the leakiness (Ki) of the BBB, brain blood volume, capillary mean transit and distribution of transit times are estimated together with brain tissue perfusion (CBF). Other functional MRI measures are obtained such as the brain microstructural organization, measured by diffusion sensitive MRI and brain activity by Blood-oxygenation level dependent Imaging and brain lactate production as a measure of brain metabolism.
4. The 360-degree evaluation of the entire project is a joint, narrative process where patients, researcher and students involved sit together using a process evaluating principle. A data triangulation and a reflection of pros and cons of the project will guide the process. The evaluation is guided by an expert in process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Post concussion syndrome (PCS) diagnose according to WHO ICD-10 classification and documented by written statement from physician veritying a mild traumatic brain injury
* Longer lasting symptoms for at least 4 weeks after initial trauma
* If allocated to add-on exercise protocol participant must feel able to prioritize the intervention structure
* Communication language must be Danish

Exclusion Criteria:

* Other diseases blurring the diagnose PCS
* Other serious brain diseases
* Severe cardiovascular diseases precluding physical activity according to protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Buffalo Concussion Bike Test from baseline measurement to week 12 | Change in Buffalo Concussion Bike Test at week 12
  Buffalo Concussion Bike Test is an individualized bike test designed to measure the number of minutes that the patient can cycle without symptom aggrevation. The test is stopped when symptoms worsen judged by VAS, BORG RPE and pulse rate. The result is measured in minutes

SECONDARY OUTCOMES:
Changes in Rivermead Post Concussion Questionaire from baseline to week 12 | Change in point score at week 12
  A systematic questionary related to patient perception of commotio during past 24 hours. Result is in point with a maximum possible score of 3 and 13 points
Changes in Fatique Scale Questionaire from baseline to week 12 | Change in point score at week 12
  A systematic questionary related to patient perception of fatique. Result is in points with a maximum possible score of 63 points
Change in Buffalo Concussion Bike Test from baseline measurement to week 4 | Change in Buffalo Concussion Bike Test at week 4
  Buffalo Concussion Bike Test is an individualized bike test designed to measure the number of minutes that the patient can cycle without symptom aggrevation. The test is stopped when symptoms worsen judged by VAS, BORG RPE and pulse rate. The result is measured in minutes
Change in Buffalo Concussion Bike Test from baseline to week 8 | Change in Buffalo Concussion Bike Test at week 8
  Buffalo Concussion Bike Test is an individualized bike test designed to measure the number of minutes that the patient can cycle without symptom aggrevation. The test is stopped when symptoms worsen judged by VAS, BORG RPE and pulse rate. The result is measured in minutes
Description of patient perspectives of living with PCS | Assessed at week 12
  In a grounded theory frame we develop new descriptions of patient experiences
Evaluation of the project | After completion of the 12 week intervention
  In a SWOT analyses frame we develop qualitative concepts of the project
Change in Sms tracking domain one: "Physical Ability" of self reported well being in relation to commotio | Change in perceived physical ability at week 12
  All included patients fill out an electronic questionary related to five domains of well being. Result of score is a number from 0 to 10
Change in Sms tracking domain two: "Overall physical symptoms" of self reported well being in relation to commotio | Change in perceived overall physical symptoms at week 12
  All included patients fill out an electronic questionary related to five domains of well being. Result of score is a number from 0 to 10
Change in Sms tracking domain three: "Using the brain" of self reported well being in relation to commotio | Change in perception of "using the brain" at week 12
  All included patients fill out an electronic questionary related to five domains of well being. Result of score is a number from 0 to 10
Change in Sms tracking domain four: "Work ability" of self reported well being in relation to commotio | Change in perception of work ability
  All included patients fill out an electronic questionary related to five domains of well being. Result of score is a number from 0 to 10
Change in Sms tracking domain five: "Quality of daily living" of self reported well being in relation to commotio | Change in perception of quality of daily life
  All included patients fill out an electronic questionary related to five domains of well being. Result of score is a number from 0 to 10
Changes in Dynamic Gait Index Questionaire from baseline to week 12 | Change in dynamic gait at week 12
  A systematic questionaire related to functional and dynamic balance during gait. Result of score is in points with a maximum of 24 points
Change in blood brain barrier permeability from baseline to week 12 | Change in blood brain barrier permeability at week 12
  Normalization of blood brain barrier permeability in the intervention group. Blood brain barrier permeability measured in mLiter/minute/mLiter of brain tissue (mL/min/mL)
Change of brain oxygen consumption from baseline to week 12 | Change of brain oxygen consumption at week 12
  Normalization of oxygen consumption in the intervention group. Measured in unit mmol oxygen/minute/ mLiter of brain tissue (mmol/min/mL).
Change of brain diffusion from baseline to week 12 | Change of brain diffusion at week 12
  Normalization of brain diffusion in the post concussion intervention patient group. Diffusion coefficient is measured in meter^2/second (m^2/s).
Change of brain lactate from baseline to week 12 | Change of brain lactate at week 12
  Normalization of lactate in the intervention group. Measurement of lactate in mmol/ml brain tissue.
Case- control comparison; Blood brain barrier permeability | Comparison measurements at baseline
  Blood brain barrier permeability measurement comparison between healthy controls and patients with post concussion syndrome. Measurement in mLiter/minute/mLiter of brain tissue (mL/min/mL)
Case-control comparison; Brain oxygen consumption | Comparison measurements at baseline
  Global brain oxygen consumption normalized to total brain volume comparison between healthy controls and patients with post concussion syndrome. Measured in unit mmol oxygen/minute/ mLiter of brain tissue (mmol/min/mL)
Case-control comparison; Brain diffusion coefficient | Comparison measurements at baseline
  Brain water diffusion coefficient comparison between healthy controls and patients with post concussion syndrome. Diffusion coefficient measured in meter^2/second (m^2/s).
Case-control comparison; Brain lactate | Comparison measurements at baseline
  Measurement of brain lactate in precuneus comparison between healthy controls and patients with post concussion syndrome. Measurement in mmol/ml brain tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik BW Larsson, Professor, Principal Investigator — Faculty of Health and Medical Science, University of Copenhagen, Denmark
Locations (1):
- University College Copenhagen, Copenhagen, Region of Greater Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No